## Janssen Research & Development \*

## **Statistical Analysis Plan (Final CSR)**

A Multicenter, Parallel-group Study of Long-term Safety and Efficacy of CNTO 136 (sirukumab) for Rheumatoid Arthritis in Subjects Completing Treatment in Studies CNTO136ARA3002 (SIRROUND-D) and CNTO136ARA3003 (SIRROUND-T)

## Protocol CNTO136ARA3004; Phase 3

## CNTO 136 (sirukumab)

\*Janssen Research & Development is a global organization that operates through different legal entities in various countries. Therefore, the legal entity acting as the sponsor for Janssen Research & Development studies may vary, such as, but not limited to Janssen Biotech, Inc.; Janssen Products, LP; Janssen Biologics, BV; Janssen-Cilag International NV; Janssen, Inc; Janssen Sciences Ireland UC; or Janssen Research & Development, LLC. The term "sponsor" is used throughout the protocol to represent these various legal entities; the sponsor is identified on the Contact Information page that accompanies the protocol.

No Statistical Analysis Plan was created for the abbreviated final Clinical Study Report for Protocol CNTO136ARA3004.

| Affirmed by: | |
|----------------------------------------|---------------------|
| | of Apr Rolq |
| Yusang Jiang, MA<br>Study Statistician | Date (Day Mon Year) |

**Status:** 

Approved

Date:

9 April 2019

Prepared by:

Janssen Research & Development, LLC; Janssen Research & Development, a division of

Janssen Pharmaceutica NV